CLINICAL TRIAL: NCT00632489
Title: A Phase I Study of LBH589 in Combination With Capecitabine ± Lapatinib
Brief Title: LBH589 in Combination With Capecitabine Plus/Minus (±) Lapatinib in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 119
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Refractory Malignancy; Breast Cancer; LBH589; Capecitabine; Lapatinib
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Panobinostat; Capecitabine; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LBH589 with Capecitabine (Experimental): MTD, LBH589 with Capecitabine
  Interventions: Drug: LBH589; Drug: Capecitabine
- LBH589 and Lapatinib (Experimental): LBH589 and Lapatinib
  Interventions: Drug: LBH589; Drug: Lapatinib
- LBH589, Capecitabine and Lapatinib (Experimental): LBH589, Capecitabine and Lapatinib (Breast Cancer Patients)
  Interventions: Drug: LBH589; Drug: Capecitabine; Drug: Lapatinib

INTERVENTIONS:
Drug: LBH589 — LBH589 will be evaluated when administered twice weekly at the following possible dose levels: 20 mg, 30 mg, 45 mg, and 60 mg. Capecitabine will be paired with LBH589 and will range in dose from 825 mg/m2 to 1250 mg/m2 orally BID 14 of every 21 days. Treatment cycles will be 21 days in length. Once determined safe, 10 additional patients will be treated at the determined MTD to further assess safety.
  Other Names: Panobinostat
Drug: Capecitabine — Capecitabine will be administered orally twice daily for 14 days out of every 21 days.
  Other Names: Xeloda
  Arms: LBH589 with Capecitabine; LBH589, Capecitabine and Lapatinib
Drug: Lapatinib — Lapatinib, 1000 mg PO daily will be added to this combination.
  Other Names: Tykerb; Tyverb
  Arms: LBH589 and Lapatinib; LBH589, Capecitabine and Lapatinib

SUMMARY:
This single center Phase I dose escalation trial will evaluate the safety, tolerability and efficacy of LBH589 when combined with capecitabine and lapatinib in three parts. Part 1 will determine the maximum tolerated doses (MTD) of LBH589 when combined with capecitabine. Parts 2 and 3 will be limited to locally recurrent or metastatic breast cancer patients, ICH 3+ overexpression or FISH amplification documented locally. Part 2 will evaluate the safety of the MTD of LBH589 determined in Part 1 when paired with lapatinib 1000 mg by mouth (PO) daily. Parts 2 and 3 will be limited to locally recurrent or metastatic breast cancer patients, ICH 3+ overexpression or FISH amplification documented locally. Part 3 will evaluate the tolerability and effectiveness of the triplet combination, LBH589, capecitabine and lapatinib in breast cancer patients.

DETAILED DESCRIPTION:
LBH589 will be evaluated when administered twice weekly at the following possible dose levels: 20 mg, 30 mg, 45 mg, and 60 mg. Capecitabine will be paired with LBH589 and will range in dose from 825 mg/m2 to 1250 mg/m2 orally BID 14 of every 21 days. Treatment cycles will be 21 days in length. Once determined safe, 10 additional patients will be treated at the determined MTD to further assess safety.

The second portion of this study will assess QTc prolongation with the LBH589 and lapatinib combination. A subset of 6 patients will be treated with the LBH589 one dose below the MTD determined during Part I. If tolerated, 6 additional patients will receive LBH589 at the MTD established in Part I with lapatinib (capecitabine will not be administered in this subset of patients).

If there are no clinically significant findings in the LBH589 and lapatinib subset, the study will advance to a third portion which combines the three drugs LBH589, capecitabine, and lapatinib.

The triple combination will initially administer lapatinib 1000 mg orally daily with LBH589 and capecitabine at one dose level below the established MTD. If tolerated, LBH589 and capecitabine doses will be escalated to the MTD.

Toxicity assessments will be ongoing and disease assessments will be repeated every 2 treatment cycles. If all dose level combinations are explored, a total of 45-55 patients will be required to accommodate for the additional patients enrolled in the QTc subset and to establish the recommended phase II dose of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented metastatic or locally unresectable, incurable malignancy for which capecitabine is clinically appropriate.
2. Male or female patients aged ≥ 18 years old.
3. Maximum of 3 prior regimens in a metastatic setting allowed and may include other targeted agents, immunotherapy and chemotherapy.
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
6. Baseline MUGA or ECHO must demonstrate LVEF > than the lower limits of the institutional normal.
7. Laboratory values as follows:

   * ANC > 1500/μL
   * Hgb > 9 g/dL
   * Platelets > 100,000/uL
   * Bilirubin < 1.5 mg/dL
   * AST/SGOT < 2.5 x ULN or < 5.0 x ULN and ALT/SGPT in patients with liver metastases
   * Creatinine < 1.5 mg/dL or calculated creatinine clearance > 50 ml/min
   * Albumin > 3 g/dL
   * Potassium > lower limit of normal (LLN)
   * Phosphorous > LLN
   * Calcium > LLN
   * Magnesium > LLN
8. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment and must commit to begin two acceptable methods of birth control, one highly effective method of birth control and one additional effective method at the same time before starting treatment.
9. Life expectancy > 12 weeks.
10. Accessible for treatment and follow-up.
11. All patients must be able to understand the nature of the study and give written informed consent prior to study entry.

Additional Breast Cancer Patient Subset (Part 2 and Part 3) Inclusion Criteria:

1. Incurable carcinoma of the breast, with measurable locally recurrent or metastatic disease.
2. ICH 3+ overexpression or FISH amplification documented by a local laboratory in primary or metastatic tumor tissue.
3. Prior treatment with an anthracycline, taxane, and trastuzumab or not a candidate for such treatment. Patient may have received these drugs in combination or in sequence for the treatment of locally advanced or metastatic disease and/or adjuvant therapy.

Exclusion Criteria:

1. Prior treatment with an HDAC inhibitor or current treatment with valproic acid.
2. Previous treatment with capecitabine.
3. Impaired cardiac function including any of the following:

   * Screening ECG with a QTc > 450 msec.
   * Congenital long QT syndrome.
   * History of sustained ventricular tachycardia.
   * Any history of ventricular fibrillation or torsades de pointes.
   * Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate > 50 beats per minute are eligible.
   * Myocardial infarction or unstable angina within 6 months of study entry.
   * Congestive heart failure (NY Heart Association class III or IV).
   * Right bundle branch block and left anterior hemiblock (bifascicular block).
   * Atrial fibrillation or flutter.
   * Ongoing therapy with antiarrhythmics or other medications associated with QTc prolongation.
4. Uncorrected hypokalemia or hypomagnesaemia.
5. Uncontrolled hypertension (systolic blood pressure [BP] 180 or diastolic BP > 100 mm Hg) or uncontrolled cardiac arrhythmias.
6. Active CNS disease, including meningeal metastases.
7. Known diagnosis of human immunodeficiency virus (HIV) infection.
8. Unresolved diarrhea > CTCAE grade 1.
9. Concomitant requirement for medication classified as CYP3A4 inducers or inhibitors.
10. Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib.
11. Patients with known hypersensitivity to 5-fluorouracil chemotherapy, investigational drug therapy, major surgery < 4 weeks prior to starting study drug or patients that have not recovered from side effects of previous therapy.
12. Patient is < 5 years free of another primary malignancy except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
13. Concomitant use of any anti-cancer therapy or radiation therapy.
14. Pregnant or breast feeding or female of reproductive potential not using two effective methods of birth control.
15. Male patients whose sexual partners are women of childbearing potential not using effective birth control.
16. Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
17. Other concurrent severe, uncontrolled infection or intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
18. Patients taking any medications listed in "Prohibited Medications" for both capecitabine and lapatinib .
19. Patients with uncontrolled coagulopathy (PT and/or PTT > 1.2 x ULN; patient must also be on stable dose of anticoagulant for a defined medical indication).
20. Abnormal thyroid function (TSH or free T4) detected at screening. Patients with known hypothyroidism who are stable on thyroid replacement are eligible.

Additional Breast Cancer Patient Subset (Part 2 and Part 3) Exclusion Criteria:

1. Prior treatment with lapatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Burris, III, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LBH589 With Capecitabine | LBH589 and Lapatinib | LBH589, Capecitabine and Lapatinib
Started | 15 | 5 | 0
Completed | 0 (Pts remained on study until disease progression, intolerable toxicity or other reason to discontinue) | 0 (Pts remained on study until disease progression, intolerable toxicity or other reason to discontinue) | 0 (Pts remained on study until disease progression, intolerable toxicity or other reason to discontinue)
Not Completed | 15 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LBH589 With Capecitabine | LBH589 and Lapatinib | LBH589, Capecitabine and Lapatinib | Total
Number analyzed (Participants) | 15 | 5 | 0 | 20
Age, Continuous [Median (Full Range); unit: years] | 54 [45 to 69] | 66 [64 to 68] |  | 56 [45 to 69]
Gender [Number; unit: participants]
  Female | 8 | 5 |  | 13
  Male | 7 | 0 |  | 7
Region of Enrollment [Number; unit: participants]
  United States | 15 | 5 |  | 20

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Maximum Tolerated Doses (MTD) and Dose-limiting Toxicities (DLT) of LBH589 in Combination With Capecitabine When Administered to Patients With Refractory and Advanced Tumor Types That Are Sensitive to 5-fluorouracil
Description: MTD for Capecitabine, BID
Time Frame: 18 months
Population: MTD Determination only for part I patients (per protocol)
Measure: Number; unit: mg/m2
Arm/Group | LBH589 With Capecitabine | LBH589 and Lapatinib | LBH589, Capecitabine and Lapatinib
Number analyzed (Participants) | 15 | 0 | 0
mg/m2 | 100 |  |

2. Secondary Outcome: To Evaluate the Antitumor Activity of LBH589 in Combination With Capecitabine in Patients With Refractory and Advanced Tumors
Time Frame: 18 months
Reporting Status: Not Posted

3. Secondary Outcome: To Evaluate the Tolerability and Preliminary Efficacy of Established Doses of LBH589 and Capecitabine With Lapatinib in a Limited Number of Patients With HER2+ Breast Cancer
Time Frame: 18 months
Reporting Status: Not Posted

4. Primary Outcome: To Determine the Maximum Tolerated Doses (MTD) and Dose-limiting Toxicities (DLT) of LBH589 in Combination With Capecitabine When Administered to Patients With Refractory and Advanced Tumor Types That Are Sensitive to 5-fluorouracil
Description: MTD for Panobinostat, twice weekly
Time Frame: 18 months
Measure: Number; unit: mg
Arm/Group | LBH589 With Capecitabine | LBH589 and Lapatinib | LBH589, Capecitabine and Lapatinib
Number analyzed (Participants) | 15 | 0 | 0
mg | 30 |  |

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | LBH589 With Capecitabine | LBH589 and Lapatinib | LBH589, Capecitabine and Lapatinib
Serious Adverse Events (participants affected / at risk) | 6/15 | 3/5 | 0/0
Other Adverse Events (participants affected / at risk) | 11/15 | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 With Capecitabine (N=15) | LBH589 and Lapatinib (N=5) | LBH589, Capecitabine and Lapatinib (N=0)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, disease progression (General disorders) | 2 | 1 | 0
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 0 | 1 | 0
Infections and infestations - Other, unspecified (Infections and infestations) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LBH589 With Capecitabine (N=15) | LBH589 and Lapatinib (N=5) | LBH589, Capecitabine and Lapatinib (N=0)
VOMITING (Gastrointestinal disorders) | 7 | 5 | 0
FATIGUE (General disorders) | 5 | 4 | 0
ANOREXIA (Metabolism and nutrition disorders) | 3 | 5 | 0
DIARRHOEA (Gastrointestinal disorders) | 5 | 3 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 5 | 0
CONSTIPATION (Gastrointestinal disorders) | 4 | 3 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 2 | 0
MUCOSAL INFLAMMATION (General disorders) | 3 | 2 | 0
DIZZINESS (Nervous system disorders) | 1 | 3 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 3 | 0
DYSPEPSIA (Gastrointestinal disorders) | 3 | 0 | 0
ASTHENIA (General disorders) | 2 | 1 | 0
WEIGHT DECREASED (Investigations) | 2 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites